CLINICAL TRIAL: NCT05191199
Title: Incidence of Erectile Dysfunction in Patients Complaining of Congenital Penile Curvature
Brief Title: Studying the Incidence of Erectile Dysfunction in Patients Complaining of Congenital Penile Curvature
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham ZAAZAA, Associate Professor, Cairo University
Other Study IDs: CongCurv&ED
Record Dates: First submitted 2021-12-05; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: To Assess Erectile Function in Patients Complaining of Congenital Penile Curvature
Keywords: Congenital penile curvature, Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal erectile response: Peak systolic velocity above 35cm/s, EDV below 5cm/s, Erectile score 4 or 3
  Interventions: Diagnostic Test: Penile Duplex Study
- Abnormal erectile response: Peak systolic velocity below 35cm/s, EDV above 5cm/s, Erectile score 2 or 1
  Interventions: Diagnostic Test: Penile Duplex Study

INTERVENTIONS:
Diagnostic Test: Penile Duplex Study — A penile duplex study will be done to assess PSV, EDV, RI, angle and degree of curvature and Erection quality using the erection hardness grading scale

SUMMARY:
Patients complaining of congenital penile curvature were subject to Penile duplex study to assess their curvature. Their penile duplex data including Peak Systolic velocity, End Diastolic velocity and Resistivity index were recorded as well as their assessing the degree of curvature and the quality of their erection using the erection hardness grading scale.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of congenital curvature

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult males
Study Population: Adult males complaining of congenital penile curvature
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Penile duplex study parameters | 3 years
  A penile duplex study will be done to assess peak systolic velocity, end diastolic velocity, Resistivity index
Degree of curvature | 3 years
  Angle and degree of penile curvature using a compass
Erection quality using the erection hardness grading scale | 3 years
  A score of 1 indicates that the penis is larger than normal, but not hard; 2 means the penis is hard, but not hard enough for penetration, 3 means the penis is hard enough for penetration but not completely hard, and 4 indicates that the penis is completely hard and fully rigid

CONTACTS AND LOCATIONS:
Overall Officials: Adham ZAAZAA, MD PhD MRCS FECSM, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Upon publishing
Access Criteria: Data will become available upon reasonable request once the manuscript has been published